CLINICAL TRIAL: NCT02568501
Title: Behavioral Economic Incentives to Improve Glycemic Control Among Adolescents and Young Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-012160
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: diabetes; adolescent; young adult; behavioral economics; financial incentives; social incentives
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily feedback (Experimental): Participants receive daily feedback from wireless glucometers that transmit data on glucose monitoring adherence.
  Interventions: Behavioral: Daily feedback
- Daily Feedback, incentives (Experimental): Participants receive daily feedback from wireless glucometers that transmit data on glucose monitoring adherence. Participants are eligible for a financial incentive if adherent.
  Interventions: Behavioral: Daily feedback; Behavioral: Financial incentive

INTERVENTIONS:
Behavioral: Daily feedback — Daily feedback on glucose levels from wireless glucometers
Behavioral: Financial incentive — Participant receive a $2 daily financial incentive framed as a loss with money allocated upfront and taken away each day of non-adherence to goal
  Arms: Daily Feedback, incentives

SUMMARY:
In this study the investigators will compare a novel approach using daily financial incentives and a tiered sponsor network to motivate adolescents and young adults with type 1 diabetes to improve glycemic control.

DETAILED DESCRIPTION:
Participants will be given daily glucose monitoring goals of ≥4 glucose checks per day with ≥1 readings within goal range (70-180 mg/dL) and provided with iHealth wireless glucometers. Half of the study participants will be randomized to the 3-month intervention arm on Way to Health. The intervention includes daily financial incentives ($60 in an account at beginning of each month with $2 daily loss if non-adherent) and a 2-level tiered sponsor network (youth select 2 people who will be notified of non-adherence after 2 and 5 consecutive days). The primary outcome will be HbA1c at 3 months compared to baseline. Secondary outcomes will include HbA1c at 6 months and the proportion of participants adherent to daily glucose monitoring goals. Exit interviews will elicit intervention feasibility and feedback from a youth perspective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes
* HbA1c of 8 or greater
* Receiving care from the Childrens Hospital of Philadelphia Diabetes Center
* English-speaking
* Owns a smartphone

Exclusion Criteria:

* New diagnosis of type 1 diabetes within past year
* Unable to provide informed consent
* Already participating in another study to improve glycemic control
* Any medical conditions that would prevent completion of the study

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c by 3 months | 3 months
  Change in HbA1c from baseline to 3 months

SECONDARY OUTCOMES:
Change in HbA1c by 6 months | 6 months
  Change in HbA1c from baseline to 6 months
Glucose Monitoring Adherence by 3 months | 3 months
  Proportion of time adherence to glucose monitoring during 3 month intervention
Glucose Monitoring Adherence by 6 months | 6 months
  Proportion of time adherence to glucose monitoring during 3 month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania; Charlene Wong, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wong CA, Miller VA, Murphy K, Small D, Ford CA, Willi SM, Feingold J, Morris A, Ha YP, Zhu J, Wang W, Patel MS. Effect of Financial Incentives on Glucose Monitoring Adherence and Glycemic Control Among Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA Pediatr. 2017 Dec 1;171(12):1176-1183. doi: 10.1001/jamapediatrics.2017.3233. PMID 29059263